CLINICAL TRIAL: NCT03108430
Title: Study of Risk Factors for Developing Inhalation Pneumonia After Inhalation
Acronym: PrevAsPI-Obs
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: RNI2016-10
Record Dates: First submitted 2017-03-31; First posted 2017-04-11 (Actual); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Inhalation Pneumonia; Risk Factor
MeSH Terms: conditions — Pneumonia, Aspiration | interventions — Risk Factors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Inhalation pneumonia
  Interventions: Other: Risk factors and incidence of IP after inhalation
- Proven inhalations
  Interventions: Other: Risk factors and incidence of IP after inhalation
- Suspected inhalations (coma + anamnesis)
  Interventions: Other: Risk factors and incidence of IP after inhalation

INTERVENTIONS:
Other: Risk factors and incidence of IP after inhalation — Calculate the annual incidence of PI, the incidence of PI in inhaled patients (in each subgroup), and analyze the risk factors by logistic regression, based on the number of patients hospitalized during the study period.

SUMMARY:
Inhalation pneumonia (PI) is common in clinical practice but is rarely studied. For example, there are no data on the incidence of pneumonia after inhalation and risk factors or protective factors to develop one since it is known that anyone who inhaled does not necessarily develop an IP. There is no data on the benefit of treating inhalation by antibiotic therapy pre-emptively although this practice is common. In this context, this observational study wishes to take stock of the situation on the subject in order to determine what actions to implement to prevent IP.

ELIGIBILITY:
Inclusion Criteria:

* In intensive care: Any intubated patient who presented:
* It is a coma with GCS ≤ 12 without VAS protection, whatever the duration
* Either a proven inhalation, defined by the presence in the VAS of gastric fluid or food
* Either a suspected inhalation, defined by the extrahospital anamnesis
* In medicine :
* Any wrong way (defined by a reflex cough when taking food)
* Coma without intubation, regardless of duration or depth

Exclusion Criteria:

* Patients with VAP

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Observation of inhalations in medicine and resuscitation and collection of data likely to influence the emergence of an IP.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-08-22 (Actual); Primary Completion 2017-08-21 (Estimated); Study Completion 2017-08-21 (Estimated)

PRIMARY OUTCOMES:
Calculate the annual incidence of PI, the incidence of PI in inhaled patients (in each subgroup), and analyze the risk factors by logistic regression, based on the number of patients hospitalized during the study period. | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France